CLINICAL TRIAL: NCT05801159
Title: An Observational Study to Determine Changes in 18F-fluoropivalate-PET During Postoperative Chemoradiotherapy for Patients With Primary Glioblastoma Multiforme
Brief Title: [18F]FPIA PET-CT in Glioblastoma Multiforme (GBM)
Acronym: FAM-GBM
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 21CX6613
Record Dates: First submitted 2023-02-07; First posted 2023-04-06 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Glioblastoma Multiforme of Brain
MeSH Terms: interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The participant will undergo a blood test to measure plasma concentrations of carnitine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Positron Emission Tomography-Computerised Tomography (PET-CT) — Injection of the 18F-fluoropivalate (18F-FPIA) radiotracer followed by a whole brain static PET-CT scan.

SUMMARY:
Glioma is the most common primary malignant brain tumour in adults and has an extremely poor prognosis. Glioblastoma is the most common subtype and its most aggressive form, with an annual incidence of 3.19 cases per 100,000.

The aim of this study is to quantify the degree of fatty acid oxidation in 20 participants diagnosed with glioblastoma multiforme (GBM) that have undergone surgical resection throughout the course of their chemotherapy and radiotherapy treatment.

The investigators hypothesise that the parameters derived from longitudinal 18F-fluoropivalate (18F-FPIA) positron emission tomography (PET) will change predictably over the course of therapy in relation to response.

DETAILED DESCRIPTION:
Twenty evaluable participants with histologically confirmed glioblastoma multiforme (GBM) following surgical resection that are due to undergo treatment with chemoradiotherapy (CRT) will be enrolled into the study. The patients invited to participate in the study will provide written informed consent, but will only undergo 18F-FPIA positron emission tomography-computerised tomography (PET-CT) imaging once they have satisfied the inclusion and exclusion criteria. Once these criteria have been satisfied, eligible participants will proceed with a 18F-FPIA PET-CT post-surgical resection/prior to CRT, mid-therapy (~4-6 weeks from the start of CRT, and at the end of CRT treatment (~10-14 weeks from the end of treatment).

All the participants that are enrolled in the study will have undergone surgical resection as part of their routine clinical care from which a tissue diagnosis will be confirmed.

On the scan date, the participants will undergo a blood test to measure plasma concentrations of carnitine. During the scan, a single dose of 18F-FPIA (maximum, 370MBq) intravenous (IV) will be administered to the participant followed by a whole brain static PET-CT scan 40 minutes post-injection.

ELIGIBILITY:
Inclusion Criteria: Patients with histologically confirmed GBM following surgical resection of their tumour and are eligible for adjuvant chemoradiation with the following characteristics will be recruited:

* Age ≥18
* World Health Organisation (WHO) performance status 0 - 2.
* If female, the subject is either post-menopausal (at least 1 year), or surgically sterilized (has had a documented bilateral oophorectomy and/or documented hysterectomy for at least 2 years), or if of childbearing potential, must have a negative urine beta human chorionic gonadotropin (beta-HCG) pregnancy test done at initial screening and on the day of tracer administration. The result of the pregnancy test must be known before administration of 18F-FPIA injection.
* The subject is able and willing to comply with study procedures, and signed and dated informed consent is obtained.
* The subject has a satisfactory medical history as judged by the investigator with no significant co-morbidities, physical examination, and vital signs findings during the screening period (from 21 days before administration).
* The subject's clinical and laboratory tests are within normal limits and/or considered clinically insignificant.

Exclusion Criteria:

* The subject has received any chemotherapy, immunotherapy, biologic therapy or investigational therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of 18F-FPIA injection.
* The subject is pregnant or lactating.
* Any other chronic illness that will or musculoskeletal condition that would not allow comfortable performance of a static PET study.
* The subject has received another investigational radioactive tracer within 1 month before administration of 18F-FPIA injection.
* Unsatisfactory renal function (epidermal growth factor receptor, eGFR<60) within 3 months of [18F]FPIA injection.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed GBM following surgical resection of their tumour and are eligible for adjuvant chemoradiation.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Impact of CRT on [18F]-FPIA-detectable fatty acid metabolism | Through study completion, an average of 4 months
  Change in the [18F]FPIA maximum standardised uptake value (SUVmax) & average standardised uptake value (SUVmean) from baseline through the post-treatment PET/CT scan.

SECONDARY OUTCOMES:
Detection of post-operative residual disease | Baseline PET/CT scan (~1-4 weeks post-surgical resection)
  [18F]FPIA SUVmax & SUVmean at baseline compared to the MRI variables (standardised uptake value (SUV) and lesion-to-grey matter ration [l/g]) measured post-operatively as per standard of care.
CRT response assessment using [18F]-FPIA PET | Through study completion, an average of 4 months
  Change in [18F]FPIA SUVmax & SUVmean in patients who ultimately show progressive disease/stable disease/partial response on standard of care imaging.

OTHER OUTCOMES:
Correlation of [18F]-FPIA uptake with available tumour genetics | Through study completion, an average of 4 months
  [18F]-FPIA SUVmax & SUVmean compared with available tumour genetics.
Correlation of [18F]-FPIA with available standard of care MRI variables | Through study completion, an average of 4 months
  Change in [18F]-FPIA SUVmax & SUVmean compared with available standard of care MRI variables (standardised uptake value (SUV) and lesion-to-grey matter ration [l/g]).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Williams, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom